CLINICAL TRIAL: NCT04876352
Title: Clinical and Brain Functional MRI Effects of a Rehabilitative Training of Upper Limb Using Immersive Virtual Reality in People With Parkinson's Disease
Brief Title: Virtual-reality for Upper Limb Rehabilitation in People With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Massimo Filippi (Other)
Responsible Party: Sponsor-Investigator, Prof. Massimo Filippi, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: GR-2018-12366005
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single-blind randomized controlled trial. 40 PD patients are randomly divided into two groups: 20 in the VR-training (experimental) and 20 in the RS-training (active comparator). The assessors are blinded to the group allocation. In addition, a group of 30 healthy age- and sex-matched control is included at baseline
Who Masked: Outcomes Assessor
Masking Description: Physiotherapist, neurologists, neuropsychologists and radiologist assessing the patients are blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR-training (Experimental): Upper limb/handwriting exercises in an immersive virtual reality setting
  Interventions: Other: Upper limb/handwriting exercises in an immersive virtual reality setting (VR-training)
- RS-training (Active Comparator): The same upper limb/handwriting exercises in a real setting
  Interventions: Other: Upper limb/handwriting exercises in a real setting (RS-training)
- Healthy subjects (Other): Age- and sex-matched healthy subjects recruited to compare clinical and fMRI characteristics at baseline.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Upper limb/handwriting exercises in an immersive virtual reality setting (VR-training) — Progressively difficult multimodal physiotherapy under the augmented visual feedback induced by the VR. Participants will wear a head-mounted display and their upper limb movements during the training will be captured by a motion tracker. Patients will perform: repetition of movements of upper limb single joints (shoulder, elbow and wrist) under the augmented visual feedback provided by the use of VR in increasingly wide range of movement; active upper limb multi-joints movements under the augmented visual feedback provided by the use of VR (following trajectories designed in the virtual space - movement involving shoulder, elbow and wrist joints) and handwriting tasks and touch screen technology usage in VR context on a tablet and a smartphone.
  30 minutes of exercises, 2 times a week, for 8 weeks.
  Arms: VR-training
Other: Upper limb/handwriting exercises in a real setting (RS-training) — Participants will perform progressively difficult multimodal physiotherapy in a real setting. Participants will be encouraged to perform their upper limb movements during the training in order to perform faster and ampler movements. They will perform: repetition of movements of upper limb single joints (shoulder, elbow and wrist) in increasingly wide range of movement under the feedback provided by therapist; active upper limb multi-joints movements under the feedback provided by the therapist (following trajectories designed on a table or on a blackboard - movements involving shoulder, elbow and wrist joints) and handwriting tasks and touch screen technology usage under the supervision of the therapist.
  30 minutes of exercises, 2 times a week, for 8 weeks.
  Arms: RS-training
Other: No intervention — Only baseline evaluations, without longitudinal assessment
  Arms: Healthy subjects

SUMMARY:
The aim of this study is to assess the effect of 8-week physiotherapy training using immersive virtual reality (VR-training) compared to a physiotherapy training performed in a real setting (RS-training) on handwriting and touch screen technology-based activities, brain functional activity and cognition in patients with Parkinson's disease (PD). Both groups will perform upper limb exercises focused at improving movement amplitude and speed during several activities such as writing and using touch screen-technology. Participants randomized to VR-training (N=20) will perform exercises under the augmented visual feedback induced by the VR aimed at stimulating movement amplitude and speed. Participants randomized to RS-training (N=20) will perform exercises in a real setting.

Before training, after training (8 weeks) and at 3-month follow-up (20 weeks), subjects with PD will undergo clinical evaluations (neurological, physiotherapy and neuropsychological) while taking their regular anti-parkinsonian drugs (on-medication state). MRI scans will be acquired at each time-point to assess brain activity reorganization during off state (MRI scans will be acquired at least 12 hours after the regular evening dopaminergic therapy administration to mitigate the pharmacological effects on neural activity). A sample of matched healthy subjects (N=30) will undergo clinical, physiotherapy, neuropsychological and MRI assessments only at study entry as a benchmark.

ELIGIBILITY:
Inclusion criteria for PD patients:

* Diagnosis of idiopathic Parkinson's disease
* H&Y scale ≤ 3 while on medication
* Age ≤ 85 years
* Right-handedness with the Edinburgh Handedness Inventory Quotient
* Right-side involvement according to H&Y and Movement Disorder Society Unified Parkinson's Disease Rating Scale III (MDS-UPDRS III)
* Handwriting difficulty defined by a score greater than or equal to 1 on item II.7 of the MDS-UPDRS
* Oral and written informed consent to study participation

Inclusion criteria for healthy controls:

* Sex-matched and age-matched with PD patients;
* Right-handed;
* Oral and written informed consent to study participation.

Exclusion criteria for PD patients:

* Mini-Mental State Examination lower than 24;
* Visual impairments that interfere with the immersive virtual environment;
* (Other) upper limb deficits impeding handwriting;
* History of (other) systemic, neurologic, psychiatric diseases, head injury and cerebrovascular alterations visible at an MRI scan;
* Family history of neurodegenerative disorders;
* History of alcohol and/or psychotropic drug abuse;
* Contraindications for MRI;
* Denied oral and written informed consent to study participation.

Exclusion criteria for healthy controls:

* Mini-Mental State Examination lower than 28;
* Visual impairments that interfere with the immersive virtual environment;
* History of systemic, neurologic, psychiatric diseases, head injury and cerebrovascular alterations visible at an MRI scan;
* History of alcohol and/or psychotropic drug abuse;
* Contraindications for MRI;
* Denied oral and written informed consent to study participation

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Letters amplitude | Baseline, after 8 weeks of training and after 3-month follow-up
  Changes in letters amplitude during a repetitive handwriting task on a writing tablet. Higher amplitude reflects a better performance. Assessment during ON medication phase

SECONDARY OUTCOMES:
Systematic Screening of Handwriting Difficulties test (SOS) | Baseline, after 8 weeks of training and after 3-month follow-up
  Systematic Screening of Handwriting Difficulties test assesses handwriting quality on a paper sheet. Patients copy 5 sentences. Handwriting quality is evaluated using five items: (i) fluency in letter formation; (ii) connections between letters; (iii) regularity of letter size; (iv) space between words; and (v) straightness of the sentence. Each item is evaluated with a score ranging from zero to two. A score of zero is given when the handwriting problem does not occur or is only present in one sentence. A score of one is given if the problem appears in two or three sentences and a score of two when the problem occurs in more than three sentences. The total SOS-score is the sum of the scores on the five criteria with a range from 0 to 10, with higher scores reflecting worse quality of handwriting. Assessment during ON medication phase.
Systematic Screening of Handwriting Difficulties test (SOS) on a tablet | Baseline, after 8 weeks of training and after 3-month follow-up
  SOS will be repeated also on a tablet with a touch-screen pen in order to assess handwriting quality on tablet. Assessment during ON medication phase.
Repetitive Prewriting task on tablet | Baseline, after 8 weeks of training and after 3-month follow-up
  Repetitive Prewriting task consists in writing specific loop figures, which reflect the essential components of writing on a tablet with a pen. Movement amplitude and speed will be recorded. Higher amplitude and speed reflect better results. Assessment during ON medication phase
Funnel task on tablet | Baseline, after 8 weeks of training and after 3-month follow-up
  Funnel task consists in alternating upstroke and down stroke writing-like movements at varying amplitudes on a tablet with a pen to assess freezing during writing. Movement amplitude and speed will be recorded. Higher amplitude and speed reflect better results, number of interruptions during writing will be recorded to assess freezing severity. Assessment during ON medication phase.
Brain functional changes during hand-tapping in a virtual reality setting | Baseline, after 8 weeks of training and after 3-month follow-up
  Changes in functional MRI brain activity assessed during hand-tapping task in a virtual reality setting. Assessment during OFF medication phase, at least 12 hours after last medication assumption.
Brain functional changes during hand-tapping in a real setting | Baseline, after 8 weeks of training and after 3-month follow-up
  Changes in functional MRI brain activity assessed during hand-tapping task in a real setting. Assessment during OFF medication phase, at least 12 hours after last medication assumption.
Hand tapping task | Baseline, after 8 weeks of training and after 3-month follow-up
  Amplitude and speed of hand tapping performed with electromagnetic sensors placed on the hand. Higher movement amplitude and speed reflect better performance. Assessment during ON medication phase.
Finger tapping task | Baseline, after 8 weeks of training and after 3-month follow-up
  Amplitude and speed of finger tapping performed with electromagnetic sensors placed on the hand. Higher movement amplitude and speed reflect better performance. Assessment during ON medication phase.
Velocity of swipe-slide finger movements on a screen | Baseline, after 8 weeks of training and after 3-month follow-up
  Velocity of swipe-slide movements of the fingers on a smartphone screen. Movements usually employed to unlock and use smartphones/tablets. Number of movements in a given time and velocity of movements reflect better performance. Assessment during ON medication phase.
Velocity of finger tapping movements on a screen | Baseline, after 8 weeks of training and after 3-month follow-up
  Velocity of tapping movements of the fingers on a smartphone screen. Movements usually employed to unlock and use smartphones/tablets. Number of movements in a given time and velocity of movements reflect better performance. Assessment during ON medication phase.
Rubber Hand Illusion paradigm | Baseline, after 8 weeks of training and after 3-month follow-up
  Rubber hand illusion assesses bodily self-awareness and sense of agency. Patients report in a 10-points level scale their agreement relatively to nine statements reflecting how is the perception of their real hand relative to the rubber hand. Higher scores reflect higher illusion. Assessment during ON medication phase.
Cambridge Neuropsychological Test Automated Battery (CANTAB) | Baseline, after 8 weeks of training and after 3-month follow-up
  This battery of cognitive tests assesses executive-attentive functions, memory and visuospatial abilities. Lower reaction time and greater number of correct responses reflect better performance. Assessment during ON medication phase.
Parkinson's Disease Questionnaire (PDQ-39) score | Baseline, after 8 weeks of training and after 3-month follow-up
  Parkinson's Disease Questionnaire investigates the quality of life of PD patients. It includes 39 questions with 5 possible answers (never, occasionally, sometimes, often, always) and 8 sub-items related to mobility, ADLs, emotional well-being, signs of discouragement, social support, cognitions, communication and bodily discomfort. The maximum score is 100 and a low score is an indicator of a good quality of life.
Manual Ability Measure (MAM-36) questionnaire | Baseline, after 8 weeks of training and after 3-month follow-up
  The Manual Ability Measurement (MAM-36) includes 36 items assessing perceived ease or difficulty in performing common tasks (e.g. eating, dressing, button clothes). Items are rated on a 4-point scale from one "I cannot do it" to four "I can do it without any problem". A zero-response option is also included, indicating tasks that are almost never performed, with or without hand impairment. Scores on the 36 items are summed to create a total score with a range from 36 to 144, with higher scores reflecting higher ability.
Purdue Pegboard Test (PPT) | Baseline, after 8 weeks of training and after 3-month follow-up
  Purdue Pegboard Test is a widely used test to assess upper limb motor function and activity. Patient is asked to place pegs vertically in a board in front of him as fast as possible for 30 seconds. Higher number of placed pegs reflects a better performance. Assessment during ON medication phase.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corbetta D, Sarasso E, Gardoni A, Zenere L, Balestrino R, Smits-Engelsman B, Pelosin E, Filippi M, Agosta F. Construct validity, intrarater and interrater reliability of the Italian version of the systematic screening of handwriting difficulties (SOS) test in people with Parkinson's disease. J Neurol. 2025 Sep 8;272(9):620. doi: 10.1007/s00415-025-13365-w. PMID 40920242